CLINICAL TRIAL: NCT07384962
Title: Prospective Evaluation of the Impact of Prior Ventral Hernia Repair on Subsequent Reoperations and Neurological Sequelae, Comparing Intra-peritoneal vs. Extra-peritoneal Mesh Placement: the ORION Study
Brief Title: ORION Study: Mesh Position and Risk During Subsequent Minimally Invasive Abdominal Surgery
Acronym: ORION
Status: Not yet recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 38X502
Record Dates: First submitted 2026-01-27; First posted 2026-02-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Ventral Hernia Repair
Keywords: ventral hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intraperitoneal mesh: This group includes adult patients who previously underwent minimally invasive ventral hernia repair with intraperitoneal mesh placement, defined as a prosthetic mesh positioned within the peritoneal cavity in direct contact with the abdominal viscera. Mesh fixation methods may include sutures, absorbable or non-absorbable tackers, glue, or mixed techniques, according to standard clinical practice at the time of the index operation.
  Patients in this group undergo subsequent minimally invasive abdominal surgery for any indication and are prospectively evaluated for intraoperative findings and postoperative outcomes, including adhesions, visceral injury during adhesiolysis, and early postoperative morbidity.
- Extraperitoneal mesh group: This group includes adult patients who previously underwent minimally invasive ventral hernia repair with extraperitoneal mesh placement, defined as a prosthetic mesh positioned outside the peritoneal cavity, either in the preperitoneal or retromuscular plane. Mesh fixation methods may include sutures, absorbable or non-absorbable tackers, glue, or mixed techniques, according to standard clinical practice at the time of the index operation.
  Patients in this group undergo subsequent minimally invasive abdominal surgery for any indication and are prospectively evaluated for intraoperative findings and postoperative outcomes, including adhesions, visceral injury during adhesiolysis, and early postoperative morbidity.

SUMMARY:
Ventral hernia repair is one of the most commonly performed abdominal surgical procedures worldwide, increasingly carried out using minimally invasive techniques. In this setting, mesh reinforcement is standard practice, but the optimal anatomical plane for mesh placement remains debated. Intraperitoneal and extraperitoneal mesh positions may have different long-term consequences, particularly when patients undergo subsequent abdominal surgery. However, prospective data evaluating the impact of prior mesh position on reoperative risk and postoperative outcomes are limited.

The ORION study is a prospective, multicentre, observational cohort study designed to evaluate the impact of prior minimally invasive ventral hernia repair with intraperitoneal versus extraperitoneal mesh placement on subsequent minimally invasive abdominal surgery. The primary objective is to compare the incidence of intraoperative visceral injury during adhesiolysis between the two mesh positions. Secondary objectives include the assessment of adhesion burden and severity, duration and extent of adhesiolysis, conversion to open surgery, and adhesion-related postoperative complications.

In a predefined subgroup of patients undergoing surgery for ventral hernia recurrence, the study also evaluates short-term postoperative outcomes, including chronic post-surgical pain, neuropathic pain features, sensory disturbances, and analgesic use.

By prospectively collecting standardized intraoperative and postoperative data across multiple centres, the ORION study aims to provide real-world evidence on the long-term surgical and functional implications of mesh positioning in minimally invasive ventral hernia repair.

ELIGIBILITY:
Inclusion Criteria

* Adults aged 18 years or older.
* Patients who previously underwent minimally invasive ventral hernia repair (primary, incisional, or recurrent) with intraperitoneal or extraperitoneal mesh placement.
* Patients scheduled to undergo elective or emergency minimally invasive abdominal surgery for any indication (including, but not limited to, hernia recurrence, bowel obstruction, cholecystectomy, colorectal, or gynecologic procedures).
* Patients in whom an initial minimally invasive approach is attempted, even if conversion to open surgery occurs after exploratory access or adhesiolysis.
* Ability to provide written informed consent, according to local regulations.

Exclusion Criteria

* Patients undergoing primary open abdominal surgery without an initial minimally invasive approach.
* Patients with a history of open ventral hernia repair as the index hernia procedure.
* Patients without available information on prior mesh position.
* Patients who decline or are unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients (≥18 years) with a history of minimally invasive ventral hernia repair involving prosthetic mesh placement, who subsequently undergo elective or emergency minimally invasive abdominal surgery for any indication. Patients are grouped according to the anatomical position of the previously implanted mesh, classified as intraperitoneal or extraperitoneal (preperitoneal or retromuscular).
  The study population is designed to reflect real-world surgical practice and includes consecutive patients undergoing a wide range of abdominal procedures, including surgery for hernia recurrence and non-hernia-related indications. Both laparoscopic and robotic approaches are eligible. In patients undergoing surgery for ventral hernia recurrence, postoperative follow-up is performed to assess early surgical, neurological, and patient-reported outcomes, while patients undergoing surgery for other indications are evaluated for intraoperative outcomes only.
Sampling Method: Probability Sample
Enrollment: 790 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of intraoperative visceral injury during adhesiolysis | During the subsequent minimally invasive abdominal surgical procedure
  The primary outcome is the occurrence of intraoperative visceral injury during adhesiolysis in patients undergoing subsequent minimally invasive abdominal surgery after previous minimally invasive ventral hernia repair. Visceral injury is defined as any unintended injury to abdominal organs, including serosal tears or full-thickness injuries of the small bowel, colon, or other intra-abdominal viscera, identified and recorded intraoperatively by the operating surgeon.
  The outcome will be compared between patients with prior intraperitoneal versus extraperitoneal mesh placement. The assessment is performed intraoperatively at the time of the subsequent surgical procedure.

IPD SHARING:
Plan to Share IPD: Undecided